CLINICAL TRIAL: NCT07336537
Title: Evaluating the Acceptability, Feasibility and Usability of Various Digital Biopsychosocial Conversational Data Collection Software in a Patient Population With Chronic Pain
Brief Title: Evaluating the Acceptability, Feasibility and Usability of Various Conversational Data Collection Software
Acronym: CADS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AugMend Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0001
Record Dates: First submitted 2025-10-21; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Mental Health Disorders; Behavioral Health Challenges; Ecological Momentary Assessment Best Practices
Keywords: Chronic Pain; Behavioral Health; Mental Health; Technology; Assessment; Data Collection; Biopsychosocial; Digital Health
MeSH Terms: conditions — Chronic Pain; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study uses a parallel group design to compare different digital biopsychosocial data collection methods in patients with chronic pain. Participants will be assigned to one of multiple study groups, each using a different approach to collect health information. Participants will remain in their assigned group throughout the study duration.
  The parallel design allows for direct comparison of acceptability, feasibility, and usability outcomes across different data collection approaches. Each group will complete the same types of assessments and provide feedback on their experience, enabling researchers to evaluate which methods work best for patients with chronic pain.
  Participants may complete study procedures either at home or at the MIT.nano Immersion Lab, depending on their assigned group and the technical requirements of their data collection method. All groups will provide comparable biopsychosocial information, but the format and platform through which this information is coll
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Digital Biopsychosocial Data Collection Software (Experimental): Participants in this arm will use digital software to provide biopsychosocial information about their chronic pain condition. The software will collect data about participants' pain experiences, physical functioning, emotional well-being, social circumstances, and other health-related factors.
  Participants may complete study procedures at home or at the MIT.nano Immersion Lab depending on the technical requirements and study protocol. They will interact with the digital platform to provide comprehensive health information and will be asked to provide feedback on their experience with the data collection method.
  This arm evaluates the acceptability (whether patients find the tool appropriate and are willing to use it), feasibility (whether it can be practically implemented in real-world settings), and usability (how easy and intuitive the tool is for patients) of the digital data collection approach.
  Interventions: Other: Digital Biopsychosocial Conversational Data Collection Software
- Control Standard Data Collection Method (Active Comparator): Participants in this arm will use a standard method to provide biopsychosocial information about their chronic pain condition. They will provide data about their pain experiences, physical functioning, emotional well-being, social circumstances, and other health-related factors using conventional data collection approaches.
  Participants may complete study procedures at home or at designated study locations depending on the study protocol. They will provide comprehensive health information through the assigned data collection method and will be asked to provide feedback on their experience.
  This arm serves as a comparison group to evaluate the acceptability (whether patients find the method appropriate and are willing to use it), feasibility (whether it can be practically implemented in real-world settings), and usability (how easy and intuitive the method is for patients) of standard data collection approaches.
  Interventions: Other: Standard Digital Questionnaire Data Collection

INTERVENTIONS:
Other: Digital Biopsychosocial Conversational Data Collection Software — This intervention involves participants interacting with digital conversational software that uses artificial intelligence and natural language processing to collect biopsychosocial health information. The software engages participants in dialogue-based interactions, asking questions about their chronic pain experience, physical functioning, emotional well-being, and social circumstances.
  The conversational interface adapts to participant responses, can ask follow-up questions for clarification, and creates an interactive experience that mimics clinical interviews. Some implementations may utilize virtual reality (VR) environments to create immersive data collection experiences at the MIT.nano Immersion Lab.
  Participants interact with the software either at home using provided devices or at the MIT.nano Immersion Lab. The AI-driven platform standardizes data collection while maintaining conversational flexibility, collecting comprehensive biopsychosocial data through natural language
  Other Names: AugMend Conversational AI Platform; Virtual Reality Biopsychosocial Data Collection Tool; CADS VR; Web CADS
  Arms: Experimental Digital Biopsychosocial Data Collection Software
Other: Standard Digital Questionnaire Data Collection — This intervention involves participants completing standard digital questionnaires or surveys to provide biopsychosocial health information. Participants respond to predetermined, fixed-format questions about their chronic pain experience, physical functioning, emotional well-being, and social circumstances.
  The data collection uses conventional electronic forms or surveys with static question sets that do not adapt based on participant responses. Questions are presented in a standard sequence without conversational elements or follow-up prompts. This represents traditional electronic data collection methods commonly used in clinical and research settings.
  Participants complete the questionnaires either at home using their own devices or provided equipment, or at designated study locations. This method provides a comparison baseline against which to evaluate newer digital data collection approaches, representing current standard practice for gathering patient-reported health informat
  Other Names: Traditional Electronic Survey Method; Static Standardized Digital Surveys
  Arms: Control Standard Data Collection Method

SUMMARY:
This research study is being conducted to evaluate digital software tools that collect health information through conversations. The study will test how acceptable, feasible, and usable these conversational software programs are for patients with chronic pain.

Purpose of the Study:

The goal is to understand whether digital conversational tools can effectively gather biopsychosocial information (biological, psychological, and social factors related to health) from patients experiencing chronic pain. Biopsychosocial information includes details about your physical symptoms, emotional well-being, social circumstances, and how these factors interact to affect your health. These digital tools are designed to have conversation-like interactions with patients to collect this comprehensive health data in a more natural and engaging way.

What Participation Involves:

If you join this study, you will interact with digital conversational software that will ask you questions about your health, pain experience, and related factors. The software is designed to communicate with you in a conversational manner, similar to talking with a healthcare provider, to gather information about your condition. You will be asked about various aspects of your chronic pain experience, including how it affects your daily life, your emotional state, and your social interactions.

Who Can Participate:

This study is looking for participants who have chronic pain conditions. Medical providers who treat patients with chronic pain are encouraged to refer eligible patients to this study. Healthcare providers interested in referring patients or learning more about the study can contact the study sponsor, AugMend Health Inc.

Why This Research Matters:

Chronic pain affects millions of people and understanding the full scope of how it impacts patients requires collecting detailed information about physical, psychological, and social factors. Traditional methods of collecting this information can be time-consuming and may not capture the complete picture. Digital conversational tools offer a potential new approach to gathering comprehensive health information in a more efficient and patient-friendly manner. This research will evaluate whether patients find these tools acceptable to use, whether they work practically in real-world clinical settings, and whether they are user-friendly and accessible for people with chronic pain.

Study Location:

The study is being conducted at AugMend Health in Cambridge, Massachusetts.

Study Sponsor:

This study is sponsored by AugMend Health Inc. Healthcare providers or potential participants who would like more information about the study or wish to make a referral can contact AugMend Health Inc.

Participation in this study is voluntary, and you can choose to stop participating at any time without affecting your regular medical care.

DETAILED DESCRIPTION:
Study Design and Methodology:

This is a research study designed to systematically evaluate various digital biopsychosocial data collection software platforms in a population of patients with chronic pain. The study will assess three key dimensions: acceptability (whether patients find the tools appropriate and are willing to use them), feasibility (whether the tools can be practically implemented in real-world clinical settings), and usability (how easy and intuitive the tools are for patients to interact with).

The study employs a comparative design to rigorously evaluate different approaches to collecting biopsychosocial information from patients with chronic pain. Participants will be assigned to use different data collection methods, allowing researchers to compare the effectiveness, user experience, and practical implementation considerations across multiple approaches. This comparative framework is essential for determining which methods work best for patients and healthcare systems.

Background and Rationale:

Chronic pain is a complex, multifaceted condition that requires comprehensive assessment of biological, psychological, and social factors to effectively understand and manage. The biopsychosocial model of pain recognizes that pain experiences cannot be fully understood by examining biological factors alone. Psychological factors such as mood, stress, coping strategies, and pain-related beliefs significantly influence pain perception and disability. Social factors including work status, family support, social isolation, and economic circumstances also play crucial roles in the chronic pain experience.

Traditional data collection methods in clinical settings often rely on paper-based questionnaires, structured interviews, or electronic forms that may not capture the nuanced, contextual information needed for holistic pain management. These conventional approaches have several limitations: they may be time-consuming for both patients and providers, can suffer from incomplete responses, may not adapt to individual patient circumstances, and often fail to capture the interconnected nature of biopsychosocial factors. Additionally, patients may experience questionnaire fatigue when faced with lengthy assessment batteries, potentially compromising data quality.

The emergence of digital health technologies has created new opportunities for patient-centered data collection. Digital platforms can potentially offer more engaging, adaptive, and comprehensive methods for gathering biopsychosocial information. However, before such tools can be widely adopted in clinical practice, it is essential to rigorously evaluate whether they meet the needs of both patients and healthcare providers. Key questions include: Do patients find these tools acceptable? Can they be practically implemented in various settings? Are they intuitive and easy for patients to use? How do they compare to existing methods?

Study Procedures and Participant Experience:

Participants enrolled in this study will engage with digital software platforms designed to collect biopsychosocial data relevant to their chronic pain condition. The software will gather information about various aspects of their pain experience, physical functioning, emotional well-being, social circumstances, and other relevant health factors.

Depending on their assigned study group, participants may interact with the data collection tools in different settings and formats. Some participants will complete study procedures at home using their own devices or equipment provided by the study team. Other participants will visit the MIT.nano Immersion Lab, a specialized research facility designed for studying human-technology interactions in controlled environments. The MIT.nano Immersion Lab provides advanced technical infrastructure and a setting specifically designed to evaluate innovative data collection approaches.

The flexibility in study locations allows researchers to evaluate how different environmental contexts may affect the data collection experience. Home-based participation offers convenience and the comfort of a familiar environment, while the laboratory setting provides controlled conditions and access to specialized equipment. Understanding how location affects acceptability, feasibility, and usability is an important aspect of determining how these tools might be deployed in real-world clinical practice.

Throughout their participation, patients will be asked to provide comprehensive feedback on their experience with the data collection methods. This feedback will help researchers understand the acceptability of the tools from the patient perspective, including factors such as comfort level with the technology, perceived relevance of the information being collected, ease of use, time required, and overall satisfaction with the experience. Participants may be asked to complete questionnaires, provide verbal feedback, or participate in debriefing sessions to share their perspectives.

Comprehensive Evaluation Framework:

The study will employ multiple methods and metrics to thoroughly evaluate the digital data collection software:

Acceptability Assessment: Researchers will evaluate whether patients find the software acceptable for collecting sensitive health information. Acceptability encompasses multiple dimensions including appropriateness (whether patients feel the method is suitable for collecting health data), comfort (whether patients feel at ease during the data collection process), willingness (whether patients are open to using this method in the future), and trust (whether patients feel confident that their information is being handled appropriately). The study will systematically document patient attitudes, preferences, concerns, and suggestions for improvement.

Acceptability may vary across different patient subgroups, and the study will examine whether factors such as age, prior technology experience, pain severity, or other characteristics influence how patients respond to the data collection methods. Understanding these variations is crucial for ensuring that new tools are accessible and acceptable to diverse patient populations.

Feasibility Assessment: The study will examine practical considerations related to implementing these tools in clinical settings and real-world environments. Feasibility assessment includes evaluating technical requirements (such as hardware, software, and internet connectivity needs), integration with existing healthcare workflows and electronic health record systems, time required for patient interactions, staff training needs, technical reliability and system stability, cost considerations, and any barriers to implementation that emerge during the study.

Feasibility is assessed from multiple perspectives including the patient viewpoint (Can patients realistically use these tools given their circumstances?), the provider perspective (Can healthcare teams incorporate these tools into their practice?), and the systems level (Can healthcare organizations successfully deploy and maintain these technologies?). The study will document technical issues, logistical challenges, and resource requirements to provide a realistic assessment of implementation feasibility.

Usability Assessment: Researchers will assess how easy the software is for patients to use and how well the design meets user needs. Usability evaluation draws on established frameworks from human-computer interaction and user experience research. Key usability dimensions include learnability (how quickly can new users understand how to use the system?), efficiency (how rapidly can users complete tasks?), memorability (can users easily use the system again after a period of not using it?), error prevention and recovery (does the system help prevent errors and allow users to recover when errors occur?), and satisfaction (how pleasant is the system to use?).

The study will identify specific usability issues that patients encounter, such as confusing instructions, unclear navigation, technical difficulties, or design elements that create frustration. This detailed feedback will inform iterative improvements to the software design. Special attention will be paid to ensuring that the tools are usable for patients with varying levels of technical proficiency and those who may have physical or cognitive limitations related to their chronic pain condition.

Population Focus and Clinical Context:

The study specifically focuses on patients with chronic pain because this population faces unique challenges in healthcare data collection and represents a significant public health concern. Chronic pain affects an estimated 20-50% of the adult population in developed countries and is one of the most common reasons for seeking medical care. The economic burden of chronic pain is substantial, including direct medical costs, lost productivity, and reduced quality of life.

Chronic pain patients often have complex medical histories involving multiple healthcare providers, various treatment approaches, and numerous medications. Many have comorbid conditions such as depression, anxiety, sleep disorders, or other chronic illnesses that interact with their pain condition. The multidimensional nature of chronic pain makes it an ideal condition for evaluating comprehensive biopsychosocial data collection tools.

Furthermore, chronic pain patients frequently interact with healthcare systems over extended periods, often for years or decades. This longitudinal nature of care makes efficient, effective, and patient-friendly data collection particularly valuable. If patients find data collection burdensome or irrelevant, engagement with care may suffer. Conversely, if data collection is perceived as valuable and manageable, it may enhance the therapeutic relationship and improve outcomes.

The chronic pain population also exhibits significant heterogeneity in terms of pain conditions (back pain, neuropathic pain, fibromyalgia, arthritis, etc.), age ranges, functional status, and psychosocial circumstances. This diversity provides an excellent opportunity to evaluate whether digital data collection tools work across different patient subgroups or whether certain approaches are better suited to specific populations.

Clinical Significance and Healthcare Impact:

The findings from this study have the potential to significantly impact how patient information is gathered in clinical settings. Current healthcare practice faces multiple challenges related to data collection: providers have limited time with patients, electronic health records are often cumbersome to use, patient-reported information may be incomplete, and the biopsychosocial factors crucial for understanding chronic conditions are frequently under-documented.

If the digital software platforms evaluated in this study prove to be acceptable, feasible, and usable for chronic pain patients, they could represent a significant advancement in healthcare data collection. Potential benefits include: reducing administrative burden on healthcare providers by automating aspects of data collection; improving the completeness and quality of patient data by using systematic collection methods; enhancing patient engagement in their own care by providing more interactive and meaningful data collection experiences; enabling more frequent monitoring of patient status between clinical visits; providing richer, more nuanced insights into the biopsychosocial factors affecting health outcomes; and creating structured data that can be more easily analyzed to identify patterns and inform treatment decisions.

Beyond chronic pain, the lessons learned from this study may have broader applicability to other chronic conditions that require comprehensive biopsychosocial assessment, such as mental health disorders, cardiovascular disease, diabetes, and cancer. The methodological approaches used in this study to evaluate acceptability, feasibility, and usability can serve as a model for assessing other digital health innovations.

Study Settings and Environmental Considerations:

The research utilizes two distinct environments to evaluate the digital data collection tools, each offering unique advantages and insights:

Home-Based Participation: Many participants will complete study procedures in their own homes. Home-based participation reflects the growing trend toward remote healthcare delivery and patient engagement outside traditional clinical settings. Evaluating tools in home environments provides ecological validity-understanding how they perform in the real-world contexts where patients actually live. Home settings may be more comfortable and convenient for patients, potentially improving participation rates and data quality. However, home environments also present challenges such as variable internet connectivity, diverse device capabilities, potential distractions, and limited technical support availability. Assessing performance in home settings helps researchers understand whether the tools are robust enough for widespread deployment.

MIT.nano Immersion Lab: Selected participants will complete study procedures at the MIT.nano Immersion Lab, a state-of-the-art facility specifically designed for studying human interactions with advanced technologies. The Immersion Lab provides controlled environmental conditions, specialized equipment, and technical infrastructure that may not be available in home or typical clinical settings. This laboratory environment allows researchers to rigorously evaluate the tools under optimal conditions and to conduct detailed assessments of user behavior and experience. The lab setting also facilitates direct observation by researchers, enabling collection of rich qualitative data about how patients interact with the technology. Additionally, the lab can accommodate equipment and technical requirements that might not be feasible for home-based deployment, allowing evaluation of more advanced or experimental approaches.

By utilizing both home and laboratory settings, the study can compare how environmental context influences the acceptability, feasibility, and usability of the data collection tools. This dual-setting approach provides a more comprehensive understanding of how the tools might perform across the spectrum of potential deployment scenarios, from controlled clinical or research environments to unstructured home settings.

Participant Safety and Ethical Considerations:

The study has received approval from WCG IRB (formerly Western Institutional Review Board), an independent ethics review board that ensures research protects participant rights, safety, and welfare. The IRB has reviewed the study protocol, consent procedures, and data protection measures to ensure they meet federal regulations and ethical standards for human subjects research.

Given that the study involves collecting sensitive health information through digital platforms, comprehensive measures are in place to protect participant privacy and ensure data security. All data collection, storage, and transmission procedures comply with applicable regulations including HIPAA (Health Insurance Portability and Accountability Act) for the protection of health information. Participants are fully informed about what information will be collected, how it will be used, who will have access to it, and how it will be protected.

Participation in this study is entirely voluntary. Patients are free to decline participation without any effect on their medical care. Those who enroll can withdraw from the study at any time, for any reason, without penalty or impact on their healthcare relationships. The informed consent process ensures that participants understand the nature of the research, what their participation involves, any potential risks or discomforts, potential benefits, alternatives to participation, and their rights as research subjects.

Data Collection and Analysis Approach:

The study will collect both quantitative and qualitative data to provide a comprehensive evaluation of the digital data collection tools. Quantitative data may include completion rates, time to complete data collection, number of technical issues encountered, standardized usability and satisfaction scores, and metrics describing the data collected. Qualitative data will include open-ended participant feedback, observations of user behavior, and detailed descriptions of implementation challenges and successes.

This mixed-methods approach allows for triangulation-using multiple data sources to develop a robust and nuanced understanding of how well the tools work. Quantitative metrics provide objective, standardizable measures that can be compared across groups and analyzed statistically. Qualitative data provides context, explanations, and insights into why certain patterns emerge and how participants experience the tools on a personal level.

Collaborative Approach and Stakeholder Engagement:

The study is designed to gather input from multiple stakeholders in the chronic pain care ecosystem. By including patients as active participants in evaluating these tools, the research ensures that the technology development is truly patient-centered and responsive to patient needs and preferences. Patient input is valued not just as data to be collected, but as expert knowledge about living with chronic pain and navigating healthcare systems.

Healthcare providers are encouraged to participate by referring eligible patients to the study. Provider involvement serves multiple purposes: it helps ensure that the study population is representative of real-world chronic pain patients seen in clinical practice; it allows providers to learn about emerging data collection approaches; and it creates opportunities for feedback about how such tools might fit into clinical workflows. Providers who refer patients can contact AugMend Health Inc. to learn more about the study and referral procedures.

The collaborative approach extends to the research team itself, which brings together expertise in chronic pain management, digital health technology, user experience research, and clinical trial methodology. This interdisciplinary collaboration ensures that the study addresses technical, clinical, and human factors considerations.

Innovation and Future Directions:

This research represents an important step in understanding how digital technologies can be applied to healthcare data collection, particularly for complex chronic conditions. The insights gained will serve multiple purposes: informing the refinement and improvement of the specific software being tested; contributing to the broader knowledge base regarding digital health tool implementation; advancing understanding of patient preferences for technology-mediated healthcare interactions; identifying best practices for biopsychosocial data collection in chronic disease populations; and informing regulatory and policy discussions about digital health tools.

The study is designed not just to answer whether specific tools work, but to generate generalizable knowledge about the factors that influence success or failure of digital health data collection tools. By systematically evaluating acceptability, feasibility, and usability, the research will identify principles and practices that can guide future innovation in this rapidly evolving field.

As healthcare increasingly incorporates digital tools and remote monitoring, understanding how to design and implement these tools effectively becomes crucial. This study contributes to that understanding by rigorously evaluating user experience, practical implementation considerations, and patient perspectives. The findings will help ensure that as healthcare adopts new technologies, these technologies truly serve the needs of patients and providers rather than creating new burdens or barriers to care.

Potential Impact on Chronic Pain Care:

Chronic pain management faces numerous challenges including limited treatment options, variability in treatment response, complex biopsychosocial contributors, and fragmented care across multiple providers. Better data collection tools have the potential to address some of these challenges by: providing clinicians with more comprehensive information about patients' pain experiences and functional status; enabling more personalized treatment planning based on detailed biopsychosocial profiles; facilitating communication between patients and providers about pain management goals and progress; supporting research to identify predictors of treatment response and develop better interventions; and empowering patients to track their own symptoms and participate more actively in their care.

While this study evaluates data collection tools rather than pain treatments per se, improvements in how pain information is gathered could indirectly lead to better pain management outcomes. Clinical decisions are only as good as the information on which they are based. If digital data collection tools can provide clinicians with richer, more accurate, and more timely information about their patients' conditions, this may translate into better treatment decisions and improved patient outcomes.

The study's focus on patient perspectives-whether patients find these tools acceptable and usable-is crucial for ensuring that any new data collection approaches will be adopted and used consistently in practice. Even the most sophisticated technology will fail if patients find it burdensome, confusing, or irrelevant. By centering patient experience in the evaluation, this research aims to identify approaches that patients will engage with willingly and consistently.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of chronic pain (pain lasting 3 months or longer)
* Able to read and understand English
* Able to provide informed consent
* Willing and able to complete study procedures either at home or at the MIT.nano Immersion Lab
* Access to necessary technology for home-based participation (if assigned to home-based group), or ability to travel to the MIT.nano Immersion Lab (if assigned to laboratory-based group)
* Cognitively able to interact with digital data collection software and provide feedback

Exclusion Criteria:

* Under 18 years of age
* Unable to provide informed consent
* Non-English speaking
* Acute pain only (pain lasting less than 3 months)
* Cognitive impairment that would prevent meaningful interaction with data collection software or ability to provide valid feedback
* Unable or unwilling to complete study procedures in assigned setting (home or laboratory)
* Any condition that, in the opinion of the investigator, would make participation unsafe or interfere with the participant's ability to complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Assessed immediately after completion of data collection procedures (typically within 1-2 weeks of enrollment)
  Acceptability will be measured using the Acceptability, Feasibility and Usability Survey (AFUS) - Acceptability Subscale, a researcher-developed instrument. This subscale includes items from Part 1 (Core Assessment Experience), Part 2 (culture), Part 3 (Future Use & Preference), Part 4 (Privacy & Trust), and Part 5 (Medical Disclosure Comfort). Items are rated on a 7-point Likert scale (1 = Strongly Disagree to 7 = Strongly Agree). Subscale scores will be calculated as the mean of all acceptability items. Higher scores indicate greater acceptability. Subscale breakdown will be accessible in supplemental figures of publications.
Usability | Assessed immediately after completion of data collection procedures (typically within 1-2 weeks of enrollment)
  Usability will be measured using the Acceptability, Feasibility and Usability Survey (AFUS) - Usability Subscale (Part 6), a researcher-developed instrument adapted from established usability frameworks. The subscale consists of 10 items rated on a 7-point Likert scale (1 = Strongly Disagree to 7 = Strongly Agree). Negatively-worded items are reverse-scored. The total score is calculated as the mean of all items. Higher scores indicate better usability.
Technical Feasibility | Assessed throughout study participation (typically within 1-2 weeks of enrollment)
  Technical feasibility will be measured by the proportion of data collection sessions completed without significant technical failures. A significant technical failure is defined as any system error, software malfunction, connectivity interruption, hardware issue, or other technical problem that results in early termination of the session. Technical success rate will be calculated as the number of sessions without significant technical failures divided by total sessions attempted, expressed as a percentage. Higher percentages indicate greater technical feasibility.
Implementation Feasibility | Assessed immediately after completion of data collection procedures (typically within 1-2 weeks of enrollment)
  Implementation feasibility will be measured using the Acceptability, Feasibility and Usability Survey (AFUS) - Future Use & Preference Subscale (Part 3). Items assess participant willingness to use the data collection method again, likelihood of recommending it to others, and trust in the method for ongoing health evaluation. Items are rated on a 7-point Likert scale (1 = Strongly Disagree to 7 = Strongly Agree). The subscale score is calculated as the mean of all items. Higher scores indicate greater implementation feasibility.
Data Collection Feasibility | Assessed at completion of all data collection procedures (typically within 1-2 weeks of enrollment)
  Feasibility of comprehensive data collection will be measured by the proportion of biopsychosocial domains for which data was successfully collected across all sessions. Domain coverage will be calculated as the number of domains with complete data divided by total possible domains, expressed as a percentage. Domains include biological (pain characteristics, sleep, physical function, nutrition), psychological (mood, cognition, coping, trauma, pain catastrophizing), and social (relationships, support, work, identity). Higher percentages indicate more comprehensive data collection.

SECONDARY OUTCOMES:
Participant Experience & Satisfaction | Assessed immediately after completion of data collection procedures (typically within 1-2 weeks of enrollment)
  Patient experience will be measured using the Acceptability, Feasibility and Usability Survey (AFUS) - Overall Experience Subscale (Part 7). Items are rated on a 7-point Likert scale (1 = Strongly Disagree to 7 = Strongly Agree). The subscale score is calculated as the mean of all items. Higher scores indicate more positive patient experience.
Patient Engagement - Session Duration | Measured during each data collection session (typically within 1-2 weeks of enrollment)
  Patient engagement will be measured by session duration, defined as the total time in minutes participants actively spend on data collection tasks, recorded via system logs. Longer durations indicate greater time engagement with the data collection process.
Patient Engagement - Response Elaboration | Measured during each data collection session (typically within 1-2 weeks of enrollment)
  Patient engagement will be measured by mean response length, defined as the average number of words per participant response across the conversation transcript. Higher word counts indicate greater verbal engagement with the data collection process. (experimental group only)
Perceived Therapeutic Alliance | Assessed immediately after completion of conversational data collection (typically within 1-2 weeks of enrollment)
  Perceived therapeutic alliance with the data collection interface will be measured using the Acceptability, Feasibility and Usability Survey (AFUS) - Therapeutic Alliance Subscale (Module A). Items are rated on a 7-point Likert scale (1 = Strongly Disagree to 7 = Strongly Agree). The subscale score is calculated as the mean of all items. Higher scores indicate stronger perceived therapeutic alliance.
Immersion and Comfort | Assessed immediately after completion of immersive data collection (typically within 1-2 weeks of enrollment)
  Immersive experience will be measured using the Acceptability, Feasibility and Usability Survey (AFUS) - Immersive Experience Subscale (Module B). Items are rated on a 7-point Likert scale (1 = Strongly Disagree to 7 = Strongly Agree). The subscale score is calculated as the mean of all items. Higher scores indicate better immersive experience.

OTHER OUTCOMES:
Correlation Between Physiological Measures and Engagement | Assessed during in-person data collection sessions (typically within 1-2 weeks of enrollment)
  The association between physiological arousal and participant engagement will be measured using correlation coefficients between Empatica-derived physiological measures (electrodermal activity, pulse rate) and engagement metrics (time spent answering questions, response word count). Correlation coefficients range from -1.0 to 1.0, with values further from zero indicating stronger associations.
Correlation Between Physiological Measures and Self-Reported Affect | Assessed during in-person study sessions (typically within 1-2 weeks of enrollment)
  The association between physiological measures and self-reported emotional states will be measured using correlation coefficients between Empatica-derived data (electrodermal activity, pulse rate, skin temperature) and participant-reported affective states from the transcripts and standardized questionnaires. Correlation coefficients range from -1.0 to 1.0, with values further from zero indicating stronger concordance between physiological and self-reported measures.
Emotive & Linguistic Analysis | Assessed at completion of the data collection (typically within 1-2 weeks of enrollment)
  Four linguistic metrics will be derived from transcripts: (1) Response Elaboration-mean words per response, with higher counts indicating greater engagement; (2) Linguistic Complexity-Flesch-Kincaid Grade Level score (0-18+) representing text sophistication; (3) Vocabulary Diversity-Type-Token Ratio (unique words/total words, 0-1.0); and (4) Self-Referential Language-percentage of first-person singular pronouns (I, me, my, mine) calculated via LIWC-22, with higher percentages associated with depression and pain catastrophizing.
Sentiment Valence of Participant Responses | Assessed at completion of the data collection (typically within 1-2 weeks of enrollment)
  Overall sentiment will be measured using automated sentiment analysis of transcripts. Sentiment scores will be calculated using validated natural language processing methods, yielding a score ranging from -1.0 (entirely negative) to +1.0 (entirely positive), with 0 representing neutral sentiment. Higher scores indicate more positive sentiment.
Thematic Content Categories | Assessed at completion of conversational data collection (typically within 1-2 weeks of enrollment)
  Thematic content of participant responses will be analyzed using qualitative thematic analysis of conversation transcripts. Two independent coders will identify recurring themes using an inductive approach, with coding disagreements resolved through consensus discussion. Inter-rater reliability will be assessed using Cohen's kappa for theme identification and reported. Results will be reported as the number of participants whose transcripts contain each identified theme (expressed as n and percentage). More prevalent themes indicate more commonly shared experiences across participants.
Topic Responsiveness | Assessed at completion of conversational data collection (typically within 1-2 weeks of enrollment)
  Participant responsiveness to questions will be measured by the percentage of questions that receive on-topic responses. Two independent coders will rate each participant response as on-topic or off-topic relative to the preceding prompt. Inter-rater reliability will be assessed using Cohen's kappa and reported. Discrepancies will be resolved through consensus discussion. Higher percentages indicate greater topic responsiveness and engagement with the structured conversation.
Disclosure Depth | Assessed at completion of conversational data collection (typically within 1-2 weeks of enrollment)
  Depth of participant self-disclosure will be measured using a researcher-developed coding scheme applied to transcripts. Two independent coders will rate each response on a 4-point scale (0 = no disclosure, 1 = factual/surface disclosure, 2 = moderate personal disclosure, 3 = deep emotional disclosure). Mean disclosure depth will be calculated across all responses. Inter-rater reliability will be assessed using intraclass correlation coefficient (ICC) and reported. Discrepancies will be resolved through consensus discussion. Higher scores indicate deeper self-disclosure.
Convergent Validity - Depression | Assessed at completion of data collection procedures (typically within 1-2 weeks of enrollment)
  Convergent validity will be assessed by comparing depression-related outputs from the data collection methods to the Patient Health Questionnaire-8 (PHQ-8). Validity will be measured using Pearson or Spearman correlation coefficients. Correlation coefficients range from -1.0 to 1.0, with values closer to 1.0 indicating stronger convergent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ruchman, MD, Principal Investigator — AugMend Health; Alexandra Therond, MA, Study Chair — AugMend Health
Locations (1):
- AugMend Health at MIT.nano Immersion Lab, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes